CLINICAL TRIAL: NCT02131649
Title: PROPS (PET/MRI Pre-Radiotherapy for Post-Prostatectomy Salvage)
Brief Title: PET/MRI for Men Being Considered for Radiotherapy for Suspected Prostate Cancer Recurrence Post-Prostatectomy
Acronym: PROPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Glenn Bauman, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GAP02-01.1
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PET; MRI; Fluorocholine; Radiotherapy; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FCH PET/MRI Scan (Experimental): Patients will undergo an injection of 18F-fluoromethyl-choline at 3.6 MBq/kg followed by whole body PET/CT imaging. Patients will also undergo a whole body MRI including T2 weighted, Diffusion weighted and Gadolinium Contrast Enhanced sequences. Patients with suspicion for recurrence may undergo biopsy if lesions identified on PET/CT or MRI are accessible for biopsy
  Interventions: Device: 18F-FCH PET/MRI Scan

INTERVENTIONS:
Device: 18F-FCH PET/MRI Scan — Patients will first undergo screening to ensure eligibility. If eligible, they will undergo a PET/MRI scan using 18F-FCH as the radiolabeled tracer. If prostate cancer is detected outside the prostate, patients may undergo a biopsy or follow-up 18F-FCH PET/MRI to confirm the results.

SUMMARY:
The PROPS trial is for men being considered for radiotherapy due to the suspicion that their prostate cancer has recurred following the surgical removal of their prostate (prostatectomy). This suspicion is based on rises seen on Prostate Specific Antigen (PSA) blood tests. Only men who demonstrate the absence of disease on standard imaging scans (Computed Tomography (CT) and bone scans) will be invited to participate.

This study will be assessing if the imaging probe 18-F Fluorocholine (18F-FCH) used during Positron Emission Tomography (PET) and Magnetic Resonance Imaging (MRI) scans, can better predict who will benefit from radiotherapy by identifying the source of cancer recurrence. This will be determined by measuring the number of men who have disease identified outside of the prostate bed (the small pocket or depression where the prostate used to be) on their 18F-FCH PET scan. Since F-18-FCH has been shown to be more sensitive in detecting prostate cancer that may have spread into lymph nodes or bone, it may potentially identify areas of prostate cancer spread not seen with standard imaging.

DETAILED DESCRIPTION:
The study will be a non-randomized, prospective study of men with suspected local recurrence of prostate cancer post-prostatectomy with negative conventional re-staging studies (bone scan and CT of the abdomen and pelvis; MRI of the pelvis as part of re-staging is allowed where it is the institutional standard of care). The clinician will develop an initial treatment plan based on conventional re-staging information.

Patients enrolled onto trial will undergo hybrid PET/MR imaging using 18F-FCH (sites without access to a hybrid PET/MR scanner will conduct a 18F-FCH PET/CT in addition to a full body MRI). A consensus staging report based on local and centralized review of the 18F-FCH PET imaging will be provided to the attending clinician, who will document a second treatment plan based on this additional information. The treatment plan to be implemented (initial or second) will be left to clinician discretion, but will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 years or older.
* Confirmation of prostate cancer on prostatectomy pathology report.
* No lymph node involvement (N0 or Nx) reported on prostatectomy pathology report.
* Documented PSA rise measured on 3 occasions.
* PSA ≥ 0.2 ng/ml at enrolment.
* At least one adverse feature: Current PSA > or equal to 1.0, Initial Gleason Grade > or equal to 8, Positive surgical margin, pT3b (seminal vesicle involvement), or PSA doubling time < 10 months.
* Bone scan and CT scan within 12 weeks of enrolment negative or equivocal for metastatic disease.
* Suitable candidate for radiotherapy and not yet had any salvage treatment post-prostatectomy.

Exclusion Criteria:

* Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components.
* Proven metastatic disease.
* Patients who refuse salvage prostate bed radiotherapy.
* Patients who refuse to join the trial or are unable to consent.
* Patients not being considered for further therapy.
* Patients who cannot lie still for at least 30 minutes or comply with imaging.
* Unequivocal evidence of disease outside the prostate bed on conventional imaging
* Allergy to MRI contrast agent (exclusion for MRI component only) or PET tracer to be used as part of the imaging
* Sickle cell disease or other anemias
* Insufficient renal function (eGFR < 30 mL/min/1.73 m2)
* Residual bladder volume > 150 cc (determined by post-void ultrasound)
* Hip prosthesis, vascular grafting or other conditions affecting imaging or delivery of therapeutic radiation
* Contraindication to MRI, including but not restricted to: pacemaker or other electronic implants, known metal in the orbit, MR incompatible surgical or cerebral aneurysm clips, Shrapnel, tattoos, non-removable body piercings (relative contraindications)
* Hormone Androgen deprivation therapy of any type within 6 months prior to enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Proportion of men with negative or equivocal conventional restaging imaging (bone scan + CT scan of abdomen and pelvis) with uptake identified outside of the prostate bed on 18F-FCH PET | Within 2 weeks of 18F-FCH PET scan

SECONDARY OUTCOMES:
Biochemical disease free survival at 3 years post-treatment | 3 years post-treatment
  Whether biochemical (PSA) control rates 3 years post-treatment are improved for participants with 18F-FCH PET imaging that was negative or demonstrated uptake confined to the prostate bed and received salvage pelvic radiotherapy compared to published results for men with adverse features.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Regional Cancer Program
Locations (10):
- Australia (4):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria
- Canada (3):
  - Lawson Health Research Institute, London Health Sciences Centre, London, Ontario
  - University of Toronto, Toronto, Ontario
  - Universite Laval Quebec, Laval, Quebec
- United Kingdom (3):
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - University College London Hospital, London
  - Royal Marsden Hospital, London